CLINICAL TRIAL: NCT02181296
Title: Effect of Local Anesthetic Concentration (0.2% Ropivacaine vs 0.1% Ropivacaine) on Phrenic Nerve Function, Pulmonary Function, and Analgesia After Ultrasound-guided Interscalene Brachial Plexus Block for Shoulder Arthroscopy
Brief Title: Pulmonary Function and Interscalene Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 820072
Record Dates: First submitted 2014-06-06; First posted 2014-07-03 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-05

CONDITIONS: Shoulder Arthroscopy
Keywords: Shoulder arthroscopy; Interscalene block; Drug concentration; 0.1% ropivacaine or 0.2% ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High concentration group (Active Comparator): 0.2% ropivacaine
  Interventions: Drug: ropivacaine
- Lower concentration group (Active Comparator): 0.1% ropivacaine
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine
  Other Names: naropin

SUMMARY:
The objective of our study is to compare the degree of phrenic nerve blockade after interscalene block using 0.1% ropivacaine or 0.2% ropivacaine. Our hypothesis is that using a lower concentration of local anesthetic will result in lesser degree of phrenic nerve block. 40 patients will be enrolled. Half will receive the block with 0.1% ropivacaine and half with 0.2% ropivacaine. Phrenic nerve and diaphragm function will be assessed by bedside spirometry and ultrasound visualization.

DETAILED DESCRIPTION:
Abstract Brief abstract (250 words or less) describing the study in language understandable to a lay person. Include brief description of the purpose, target disease/condition if applicable, key eligibility criteria, and main study interventions.

The interscalene brachial plexus block is well-suited for surgical procedures of the shoulder and proximal humerus. A well-established hazard of the interscalene block is ipsilateral hemidiaphragm paresis in nearly 100% of patients secondary to phrenic nerve blockade. This side effect is well-tolerated in most patients; however, extreme caution should be employed in patients with pulmonary disease, who may experience acute pulmonary failure from unilateral phrenic nerve blockade and resulting hemidiaphragm paresis. This study seeks to determine if using a lower concentration of ropivacaine will result in less diaphragm dysfunction and reduction in pulmonary function than a higher concentration of the local anesthetic. Patients will be randomized to one of two groups--Group A and Group B. Group A will receive ultrasound-guided interscalene block with 20mL 0.1% ropivacaine in the preoperative holding area prior to induction of general anesthesia. Group B will receive ultrasound-guided interscalene block with 20mL 0.2% ropivacaine in the preoperative holding area prior to induction of general anesthesia. The primary outcome variable is the degree of phrenic nerve blockade as assessed by ultrasonographic evaluation of diaphragm function and bedside spirometry (lung function testing). Secondary outcome variables will be assessed at various time intervals. They include oxygen saturation measurements, oxygen requirements, motor strength and sensation of blocked extremity, pain scores, opioid requirements, PACU (Post-Anesthesia Care Unit)length of stay, and patient satisfaction and quality of recovery scores. We hypothesize that interscalene brachial plexus blocks performed with a lower concentration of ropivacaine will result in less pulmonary dysfunction without compromising analgesia.

Objectives Overall objectives

1. Primary Objective: Compare the degree of phrenic nerve blockade after ultrasound-guided interscalene block using either 0.1% ropivacaine or 0.2% ropivacaine
2. Hypothesis: Using a lower concentration of local anesthetic will result in lesser degree of phrenic nerve blockade. Specifically, we hypothesize that outcome measures will be as follows for patients receiving lower concentrations of ropivacaine: 1. Less dysfunction of diaphragm movement, 2. PFT (Pulmonary Function Test) values drop less in lower concentration groups, 3. Less oxygen desaturation in PACU, 4. Less symptomatic shortness of breath post-block, 5. Less need for supplemental oxygen in PACU, 6. Less unplanned hospital admission
3. Secondary Objective: Compare the analgesia efficacy as well as block duration between 0.1% and 0.2% ropivacaine. Assess the quality of recovery as well as overall satisfaction of patients undergoing arthroscopic shoulder surgery under combined regional/ general anesthesia. Also compare and evaluate the presence of other complications that arise in the two groups Primary outcome variable(s) The primary outcome variable is the degree of phrenic nerve blockade as assessed by ultrasonographic evaluation of diaphragm function and bedside spirometry.

Secondary outcome variable(s) Secondary outcome variables include oxygen saturation measurements and oxygen requirements before block performance, 20 minutes after block performance, and in the PACU; motor strength and sensation of affected extremity before block performance, 20 minutes after block performance, and in the PACU; pain scores and opioid requirements in the PACU and up to 72 hours post-operatively, PACU length of stay, patient satisfaction and quality of recovery scores 24 hours post-operatively.

Background Describe succinctly and clearly the past findings which justify the plan for this project. A summary of the relevant literature in the area of interest and reports of previous studies should be included.

The brachial plexus, formed by the anterior roots of the spinal nerves C5- T1 innervates the shoulder, axilla, and upper extremity. The roots each exit posterior to the vertebral artery and travel laterally in the troughs of the corresponding cervical transverse processes and finally join to form trunks in the posterior cervical triangle between the anterior and middle scalene muscles. C5 and C6 join to form the superior trunk. C7 forms the middle trunk, and C8 and T1 join to form the inferior trunk. The trunks pass over the first rib and under the clavicle in association with the subclavian artery and branch into anterior and posterior divisions. The posterior divisions join to form the posterior cord. The lateral cord is formed by the anterior divisions of the superior and middle trunks. The medial cord is formed by the anterior division of the inferior trunk. The cords descend into the axilla where each has one major branch in addition to several minor branches before becoming a terminal nerve of the upper extremity. Branches of the lateral and medial cord form the median nerve. A branch off the lateral cord becomes the musculocutaneous nerve. The posterior cord becomes the radial nerve and the axillary nerve. The medial cord forms the ulnar nerve as well as the medial brachial and medial antebrachial cutaneous nerves (1,2). Each peripheral nerve has its own predictable cutaneous innervation pattern which can be mapped along the upper extremity; furthermore knowledge of peripheral nerve and dermatomal innervation can help guide decisions on which regional anesthetic approach to employ for a given surgical intervention.

The brachial plexus provides all of the motor and most of the sensory innervation to the shoulder except for the most cephalad cutaneous portion of the shoulder which receives sensory innervation from the supraclavicular nerves of the superficial cervical plexus, nerve roots C3-C4. It is therefore easy to understand that complete surgical anesthesia of the shoulder must employ a regional technique that blocks both the cervical and the brachial plexuses.

The brachial plexus can be blocked along multiple anatomic levels depending on which area of the upper extremity the procedurist wishes to anesthetize. The preferred approach depends on the surgical site and the risk of complications. The interscalene brachial plexus block is well-suited for surgical procedures of the shoulder and proximal humerus as it blocks the cervical plexus (formed by the ventral rami of C1 through C4 spinal nerve roots) in addition to the brachial plexus, effectively anesthetizing the skin of the shoulder. It is less suited for surgery of the forearm or hand as incomplete blockade of the inferior trunk results in incomplete analgesia of ulnar nerve distribution. A well-established hazard of the interscalene block is ipsilateral hemidiaphragm paresis in nearly 100% of patients secondary to phrenic nerve blockade from spread of local anesthetic around anterior scalene muscle. This side effect is well-tolerated in the majority of patients; however extreme caution should be employed in patients with COPD (Chronic Obstructive Pulmonary Disease) or other pulmonary disease, who may experience acute pulmonary failure from unilateral phrenic nerve blockade and resulting hemidiaphragm paresis. Because the interscalene nerve block provides excellent post-operative pain control for shoulder surgery and may preclude the use of general endotracheal anesthesia which has its own inherent risks in patients with severe pulmonary disease, it would be helpful to establish variables in regional technique that affect phrenic nerve blockade.

There are a few publications analyzing the degree of phrenic nerve blockade and diaphragmatic function after interscalene brachial plexus block. A detailed review of these studies has shown that both reduction in volume and concentration of local anesthetic are associated with decreased reduction in pulmonary function tests and diaphragmatic dysfunction (3,4). There are; however, still essential questions that remain unclear and improvements in study design that can be made. Specifically, the study done by Al-Kaisy et al. in 1999 which showed that lower concentrations of bupivacaine are associated with less reduction in pulmonary function and less diaphragmatic dysfunction looked at only 11 healthy volunteers. These volunteers did not have surgery after receiving blocks and therefore are not representative of a true clinical situation. In addition, the sample size of 11 is too small to draw a conclusion. Furthermore, this study used a nerve stimulator-based approach to interscalene brachial plexus blockade and therefore deposition of local anesthetic was not visualized. Without direct visualization of local anesthetic deposition, it is impossible to say that all blocks in this study were consistently performed. This lack of consistency between blocks could contribute to variance in outcomes. An ultrasound-guided block approach is more effective at maintaining consistency in block performance and may decrease variance in outcomes. Also Al-Kaisy et al. used bupivacaine and our study will be using ropivacaine (3).

All subjects enrolled in this research study are not considered to receive suboptimal treatment. The standard of care for shoulder surgery is general anesthesia plus regional anesthesia if regional anesthesia is not contraindicated. Regional anesthetics are performed with different local anesthetics of different concentrations. In fact, if our study shows that a lower concentration of ropivacaine achieves the same analgesic effect with less diaphragmatic dysfunction, many more patients who were previously deemed to not be candidates for interscalene blockade due to pulmonary disease, may receive the block and receive superior post-operative pain control than they would have had without the block.

Study Design Phase* Not applicable

Design This study is a prospective, randomized, double blinded study with 40 patients. Patients will be randomized to one of two groups--Group A and Group B. Group A will receive interscalene block with 20mL 0.1% ropivacaine in the preoperative holding area prior to induction of general anesthesia and Group B will receive interscalene block with 20mL 0.2% ropivacaine in the preoperative holding area prior to induction of general anesthesia. Interscalene blocks will be performed under ultrasound guidance by attending anesthesiologists who are experienced in regional anesthesia or by resident physicians under the direct supervision of attending anesthesiologists with experience in regional anesthesia. They will be performed in accordance with standard procedure at Penn Presbyterian Medical Center and ambulatory surgery center. The syringes of both concentrations of ropivacaine will be supplied by the research investigational pharmacy.

Study duration We plan to begin enrollment in March 2014. The enrollment of all subjects is projected to be completed in December 2014 with data analysis to follow. The study is expected to be completed by June 2015. The length of participation for each subject will be up to 72 hours in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled for shoulder arthroscopy
2. ASA physical status between I-III
3. Mentally competent and able to give consent for enrollment in the study -

Exclusion Criteria:

1. Patients who are coagulopathic or currently on anticoagulation medication (except for ASA (acetylsalicylic acid) or NSAIDS)
2. Patients with severe pulmonary disease such as asthma or COPD or substantial smoking history suggestive of COPD
3. Patients with allergy to local anesthetics or other study drugs
4. Patients with chronic opiate use
5. Patients with known dysfunction of diaphragm, intercostal muscles, or other neuromuscular disorders affecting respiration
6. Inability to speak or understand English language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Elkassabany, MD, Principal Investigator — University of Pennsylvania, Anesthesia

REFERENCES:
- [Derived] Wong AK, Keeney LG, Chen L, Williams R, Liu J, Elkassabany NM. Effect of Local Anesthetic Concentration (0.2% vs 0.1% Ropivacaine) on Pulmonary Function, and Analgesia After Ultrasound-Guided Interscalene Brachial Plexus Block: A Randomized Controlled Study. Pain Med. 2016 Dec;17(12):2397-2403. doi: 10.1093/pm/pnw057. Epub 2016 Apr 13. PMID 28025374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing shoulder arthroscopy for rotator cuff repair were recruited from the orthopedic clinic of the University of Pennsylvania.
Groups:
- High Concentration Group: 0.2% ropivacaine
  ropivacaine
- Lower Concentration Group: 0.1% ropivacaine
  ropivacaine
Period: Overall Study
Arm/Group | High Concentration Group | Lower Concentration Group
Started | 25 | 25
Completed | 18 | 19
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Concentration Group | Lower Concentration Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (15.8) | 48.3 (14.7) | 44.4 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 19 | 15 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Paradoxical Diaphragmatic Movement
Description: The primary outcome variable is the number of patients with paradoxical diaphragmatic movement ( as an indication for phrenic nerve blockade) as assessed by ultrasonographic evaluation of diaphragm
Time Frame: 30 minutes after the block
Population: Paradoxical diaphragm movement at 30 min after the block. we had missing data on 3 patients ( 2 from the 0.1% group and 1 from the 0.2% group)
Measure: Count of Participants; unit: Participants
Arm/Group | High Concentration Group | Lower Concentration Group
Number analyzed (Participants) | 24 | 23
Participants | 16 | 8

2. Secondary Outcome: Percentage Change of Forced Vital Capacity (FVC) From Pre-block Value to Value Measures in PACU
Description: The percentage change in the FVC from preblock value to values measured in PACU. The negative value represents the decrease in the FVC value.
Time Frame: within 30 minutes from arrival to PACU
Population: FVC measured within 30 minutes from arrival to PACU. We had missing data on three patients ( 2 in the 0.1% ropivacaine and 1 from the 0.2% ropivacaine group)
Measure: Median (Inter-Quartile Range); unit: percentage of change in FVC
Arm/Group | High Concentration Group | Lower Concentration Group
Number analyzed (Participants) | 24 | 23
percentage of change in FVC | -33.4 [-38 to -16] | -22 [-31.1 to -5]

3. Secondary Outcome: Percentage Change in Forced Expired Volume in First Second (FEV1) After the Block
Description: FEV1 was measured within 30 minutes of arrival to PACU. The outcomes represent the percentage change from the preoperative value to the value measured in PACU (Post-Anesthesia Care Unit). The negative value represents the decrease in the FEV1 value.
Time Frame: within 30 minutes from arrival to PACU
Population: participants post-block within 30 minutes from arrival to PACU. we had three patients with missing data on these value and hence the discrepancy between the number of patients enrolled and the number of patients analyzed ( 2 patient from the 0.1% group had missing data and one patient from the 0.2% had missing data)
Measure: Median (Inter-Quartile Range); unit: Percentage of change of FEV1
Arm/Group | High Concentration Group | Lower Concentration Group
Number analyzed (Participants) | 24 | 23
Percentage of change of FEV1 | -28 [-40 to -13] | -20 [-29 to -8]

4. Secondary Outcome: Opioid Requirements for 72 Hours After Surgery
Description: in the milligram equivalent of codeine, using web-based opioid dose converter
Time Frame: 72 hours
Population: used nonparametric test to compare between the two groups. the discrepancy of the number of patients analyzed and participants have been previously explained
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | High Concentration Group | Lower Concentration Group
Number analyzed (Participants) | 24 | 23
milligrams | 55 [25 to 75] | 102 [65 to 150]

ADVERSE EVENTS:
Time Frame: From consent to 72hrs post op
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | High Concentration Group | Lower Concentration Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No